CLINICAL TRIAL: NCT01588704
Title: A Phase II Study of Neoadjuvant Pemetrexed, Carboplatin and Bevacizumab in Unresectable, Locally Advanced Lung Adenocarcinoma
Brief Title: Neoadjuvant Pemetrexed, Carboplatin and Bevacizumab in Unresectable, Locally Advanced Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Si-Yu Wang (Other)
Responsible Party: Sponsor-Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1001; wsy002 (Other: Guangdong Province Association Study of Thoracic Oncology)
Record Dates: First submitted 2012-04-25; First posted 2012-05-01 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Lung Cancer
Keywords: lung cancer; lung adenocarcinoma; bevacizumab; adjuvant chemotherapy; surgical resection rate; safety; feasibility
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung | interventions — Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Bevacizumab (Experimental): Four cycles of neoadjuvant chemotherapy with pemetrexed, carboplatin and bevacizumab.
  Interventions: Drug: Neoadjuvant Bevacizumab

INTERVENTIONS:
Drug: Neoadjuvant Bevacizumab — Neoadjuvant Pemetrexed, Carboplatin and Bevacizumab followed by surgical resection
  Other Names: Pemetrexed (Alimta); Bevacizumab (Avastin)

SUMMARY:
The prognosis of patients with unresectable, locally advanced non-small cell lung cancer (NSCLC) is poor. Chemoradiotherapy is the main treatment modality for this disease. The newer drug regimens can be expected to improve survival in this subset of NSCLC patients. Modern targeted therapies have enhanced the outcomes of lung cancer treatment, especially for advanced NSCLC. Among the targeted approaches for the inhibition of angiogenesis is bevacizumab, a monoclonal antibody that represses vascular endothelial growth factor (VEGF). Bevacizumab in combination with platinum-based chemotherapy used as neoadjuvant chemotherapy may change the previous treatment modality. It allows some lung cancer patients to be downstaged to surgery rather than radiotherapy. Thus, survival of these patients may be improved.

DETAILED DESCRIPTION:
This trial investigates the role of neoadjuvant pemetrexed, carboplatin and bevacizumab in unresectable, locally advanced lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable, locally advanced (III A (bulky N2), III B) lung adenocarcinoma
* No previous chemotherapy, radiotherapy, surgery or biological therapy for lung cancer
* Adequate organ and bone marrow function

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for NSCLC
* Prior treatment with bevacizumab or other agents specifically targeting vascular endothelial growth factor (VEGF)
* Patients with known hypersensitivity to other recombinant human antibodies
* History of stroke or transient ischemic attack (TIA).
* History of myocardial infarction or unstable angina within the past 12 months.
* Other serious illness or medical condition including unstable cardiac disease requiring treatment, history of significant neurologic or psychiatric disorders (including psychotic disorders, dementia, or seizures), symptomatic diverticulitis, or active uncontrolled infection.
* Women who are pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Resectability rate | 3 months

SECONDARY OUTCOMES:
Number of participants with perioperative complications | 4 months
Disease-free survival | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China